CLINICAL TRIAL: NCT05133245
Title: PHACE - Prospective Genetic Investigation
Acronym: PHACE
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Karen Joos, Primary Investigator, Vanderbilt University Medical Center
Other Study IDs: 211300
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: PHACE Syndrome
MeSH Terms: conditions — Aortic Aneurysm, Giant Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic study only — Diagnostic study only

SUMMARY:
Investigation for potential PHACE syndrome gene.

DETAILED DESCRIPTION:
Subjects with PHACE syndrome diagnosis will undergo a brief physical examination with possible external photographs. Cheek swabs will be sent for genetic analysis. Subjects will be notified of the results.

ELIGIBILITY:
Inclusion Criteria:

* PHACE syndrome diagnosis
* Must be willing to have an eye examination
* Must be willing to undergo genetic testing

Exclusion Criteria:

* No PHACE syndrome diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All age groups, genders, and ethnicities who qualify with the PHACE syndrome diagnosis and consent to undergo an examination and genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Potential PHACE Gene Identification | 3 years
  Evaluation for potential PHACE gene

CONTACTS AND LOCATIONS:
Overall Officials: Karen Joos, MD, PhD, Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided